CLINICAL TRIAL: NCT00555893
Title: Monitoring Influenza Severity on Tamiflu (MIST)
Brief Title: Efficacy Study of Early Versus Late Oseltamivir Administration for Treating and Preventing Influenza
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marshfield Clinic Research Foundation (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Principal Investigator, Edward Belongia, Senior Research Scientist, Director Epidemiology Research Center, Marshfield Clinic Research Foundation, Marshfield Clinic Research Foundation
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1U01IP000124-01 (NIH)
Record Dates: First submitted 2007-11-07; First posted 2007-11-09 (Estimated); Results first posted 2015-01-14 (Estimated); Last update posted 2018-10-16 (Actual); Status verified 2018-10

CONDITIONS: Influenza
Keywords: randomized; blinded; controlled; efficacy
MeSH Terms: conditions — Influenza, Human | interventions — Oseltamivir

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active Drug (Experimental): Adults and adolescents weighing greater than 88 pounds will receive one 75 mg oseltamivir capsule twice daily, with or without food for a total of 5 days (10 doses). Participants one year of age and older up to a maximum weight of 88 pounds will receive a liquid form of study medication containing oseltamivir at a concentration of 15mg/ml. The dose will be based on weight:
  for weight <=33 lbs, dose=30 mg, volume per dose (15mg/mL)=2 mL two times per day x 5 days (10 doses); for weight 34-51 lbs, dose=45 mg, volume per dose (15mg/mL)=3 mL two times per day x 5 days (10 doses); for weight 52-88 lbs, dose=60 mg, volume per dose (15mg/mL)= 4 mL two times per day x 5 days (10 doses)
  Interventions: Drug: Oseltamivir
- Placebo (Placebo Comparator): Identical placebo capsule twice daily for 5 days (10 doses). Participants one year of age and older up to a maximum of 88 pounds will receive a placebo syrup. The dose will be based on weight as follows: <=33 pounds,2 mL doses, two times per day; 34 - 51 pounds, 3 mL doses, two times per day; 52-88 pounds, 4 mL doses, two times per day.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Oseltamivir — Adults and adolescents weighing greater than 88 pounds will receive one 75 mg oseltamivir capsule twice daily, with or without food for a total of 5 days (10 doses). Participants one year of age and older up to a maximum weight of 88 pounds will receive a liquid form of study medication containing oseltamivir at a concentration of 15mg/ml. The dose will be based on weight:
  for weight <=33 lbs, dose=30 mg, volume per dose (15mg/mL)=2 mL two times per day x 5 days (10 doses); for weight 34-51 lbs, dose=45 mg, volume per dose (15mg/mL)=3 mL two times per day x 5 days (10 doses); for weight 52-88 lbs, dose=60 mg, volume per dose (15mg/mL)= 4 mL two times per day x 5 days (10 doses)
  Other Names: Tamiflu
  Arms: Active Drug
Drug: Placebo — Identical placebo capsule twice daily for 5 days (10 doses). Participants one year of age and older up to a maximum of 88 pounds will receive a placebo syrup. The dose will be based on weight as follows: <=33 pounds,2 mL doses, two times per day; 34 - 51 pounds, 3 mL doses, two times per day; 52-88 pounds, 4 mL doses, two times per day.
  Arms: Placebo

SUMMARY:
This study is a randomized, blinded, placebo-controlled clinical efficacy trial to assess the duration and severity of influenza symptoms, and duration of viral shedding, in influenza patients receiving oseltamivir early and late relative to placebo.

There are two main hypotheses in this study:

1. The duration of influenza symptoms, mean severity score, and duration of viral shedding are reduced in patients who initiate oseltamivir treatment late (48 to 119 hours) compared to those receiving no antiviral therapy.
2. Prior influenza vaccination (same season) reduces the duration of influenza symptoms and mean symptom severity in patients receiving oseltamivir after adjusting for age and timing of antiviral therapy (early versus late).

There are two secondary hypotheses:

1. The duration of influenza symptoms, mean severity score, and duration of viral shedding are reduced in patients with influenza who initiate oseltamivir treatment early (< 48 hours) versus late (48 to 119 hours).
2. The incidence of secondary complications is lower in patients initiating oseltamivir therapy late relative to those receiving no antiviral therapy.

DETAILED DESCRIPTION:
In the past decade influenza has become increasingly recognized as a serious disease and pandemic threat. Elderly persons, young children, and individuals with chronic medical conditions have the greatest risk for complications or death from influenza infection. Neuraminidase inhibitors are currently licensed for the treatment and prevention of influenza if started early in the course of illness, but little is known regarding the effects of oseltamivir (one neuraminidase inhibitor) on illness severity when initiated later in the course of illness. Greater knowledge of the treatment effects is urgently needed for optimal management of seasonal influenza, and to maximize use of a limited stockpile of antiviral drugs in the event of an influenza pandemic.

ELIGIBILITY:
Inclusion criteria:

1. Outpatient or inpatient encounter for acute respiratory illness less than 5 days (120 hours) duration.
2. Acute respiratory illness with feverishness OR cough.
3. Access to the internet or telephone at home. This is required because symptom severity reports will be submitted twice daily using either a secure web-based form or automated telephone entry. All phones in the Marshfield area have touchtone service, allowing automated data entry.

Exclusion criteria:

1. Institutional resident (including assisted living or skilled nursing facility).
2. Self-reported chronic liver or kidney disease. These conditions are listed as precautions in the oseltamivir manufacturer package insert (www.rocheusa.com/products/tamiflu/pi.pdf).
3. Pregnancy or breast-feeding. Oseltamivir is classified as pregnancy category C, and it is excreted in breast milk. The package insert states that the drug should be used only if the potential benefit justifies the potential risk to the fetus or breast-fed infant.
4. Prior hypersensitivity reaction to oseltamivir.
5. Dementia, impaired communication, or other reason for inability to provide informed consent.
6. Immunocompromised status, including HIV infection, neutropenia, systemic corticosteroid use, or use of other immunosuppressive drugs in the past 30 days. The manufacturer states that the efficacy of oseltamivir has not been established in immunocompromised patients.
7. Patient received 1 or more doses of influenza antiviral agents (oseltamivir, zanamivir, amantadine, rimantadine) or a prescription for one of these drugs prior to randomization.

Ages: 1 Year to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 194 (Actual)
Dates: Start 2008-01; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edward Belongia, MD, Principal Investigator — Marshfield Clinic Research Foundation
Locations (1):
- Marshfield Clinic Research Foundation, Marshfield, Wisconsin, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One participant in the 194 enrolled was negative for influenza by polymerase chain reaction at randomization and was therefore excluded leaving 193 individuals started in the study.
Period: Overall Study
Arm/Group | Active Drug | Placebo
Started | 130 | 63
Final Analysis | 114 (n=16 excluded from number started because >119 hrs) | 51 (n=12 excluded from number started because >119 hrs)
Completed | 130 | 63
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Drug | Placebo | Total
Number analyzed (Participants) | 114 | 51 | 165
Age, Customized [Number; unit: years]
  <2 years | 4 | 1 | 5
  2-18 years | 54 | 28 | 82
  >18 years | 56 | 22 | 78
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65 | 34 | 99
  Male | 49 | 17 | 66
Region of Enrollment [Number; unit: participants]
  United States | 114 | 51 | 165
Influenza Type [Number; unit: participants] — Number of individuals positive by polymerase chain reaction (PCR) assay by flu type; 1 excluded who was positive for both A & B
  participants
    Type A | 85 | 38 | 123
    Type B | 28 | 13 | 41

OUTCOME MEASURES:

1. Primary Outcome: Duration of Influenza Illness
Description: Resolution is defined as occurring at the start of the first 24-hour period in which the total symptom score was less than or equal to 2 with no symptom rated higher than mild. Time to resolution was calculated from the time of randomization to symptom resolution in 12 hour increments.
Time Frame: Interval (in 12 hour blocks) from time of randomization until resolution (minimum 7 days, maximum 14 days)
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Active Drug | Placebo
Number analyzed (Participants) | 114 | 51
days | 4 [3.5 to 5] | 4 [3.5 to 4.5]

2. Secondary Outcome: Mean Illness Severity Score
Description: Mean severity score will be calculated by first summing the symptom severity scores for all reporting periods from initial enrollment (randomization) up to (and including) the first period of symptom resolution, as defined above. The summed total will be divided by the number of reporting periods to yield the mean severity score for each participant. For each reporting period, the possible symptom scores will range from 0 (all symptoms absent) to 24 (all symptoms severe). For children less than 2 years old, the possible scores will range from 0 to 15.
Time Frame: Calculated from initial enrollment (randomization) up to first period of symptom resolution (minimum of 7 days, maximum of 14 days)
Population: All participants over 24 months of age (n=5 were excluded because <24 months)
Measure: Median (Inter-Quartile Range); unit: mean severity score
Arm/Group | Active Drug | Placebo
Number analyzed (Participants) | 110 | 50
mean severity score | 6.1 [5.0 to 7.7] | 5.8 [4.8 to 7.7]

3. Secondary Outcome: Viral Shedding on Day 3-4 of Treatment
Description: Proportion of participants with positive PCR on day 3-4 of treatment
Time Frame: 3-4 days after treatment initiation
Population: 134 subjects were randomized and initiated treatment 48-119 hours after illness onset (late treatment group). Of these 95 received oseltamivir and 39 received placebo.
Measure: Count of Participants; unit: Participants
Arm/Group | Active Drug | Placebo
Number analyzed (Participants) | 95 | 39
Participants | 12 | 4

4. Secondary Outcome: Secondary Complications (Otitis Media, Sinusitis, Pneumonia, Hospital Admission)
Time Frame: 30 days from symptom onset
Population: These data were not collected because study was terminated early and did not achieve target enrollment.
Arm/Group | Active Drug | Placebo
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Mean Influenza Well-being Score
Description: Mean influenza wellbeing score is calculated by first summing the daily scores for overall health (0-9 points), ability to perform usual activities (0-9 points), and sleep quality (0-9 points) from initial enrollment (randomization) up to (and including) the first day of symptom resolution. This is divided by the number of reporting days to yield the mean daily influenza wellbeing score for each person. Minimum score is 0 and maximum is 27. Higher scores indicate better outcome.
Time Frame: Randomization to resolution
Population: The analysis is restricted to subjects randomized 48 to 119 hours after illness onset.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active Drug | Placebo
Number analyzed (Participants) | 91 | 38
score on a scale | 19.54 (3.22) | 20.04 (2.89)

ADVERSE EVENTS:
Arm/Group | Active Drug | Placebo
Serious Adverse Events (participants affected / at risk) | 0/114 | 0/51
Other Adverse Events (participants affected / at risk) | 0/114 | 0/51

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No